CLINICAL TRIAL: NCT06696586
Title: Comparison Between Effect of Systemic Fentanyl Infusion and Fentanyl Added as An Adjuvant to Lidocaine in Bier Block For Controlling Pain in Patients Undergoing Hand Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mostafa Ibrahim, resident doctor at Anaesthesia and ICU department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fentanyl Bier Block
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Bier Block; Hand Surgery
Keywords: Systemic Fentanyl Infusion; Fentanyl Added as An Adjuvant to Lidocaine
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients will be randomly allocated to one of two groups; each group consisted of 42 patients. Randomization will be performed using a closed envelope method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Experimental): patients will received lidocaine with dose 250 mg and fentanyl infusion in dose of 200 µg in rate 10ml /hr using 50ml syringe pump
  Interventions: Drug: Fentanyl infusion
- group 2 (Experimental): patients will receive lidocaine 250 mg in addition to fentanyl injection in dose 100 µg by shots
  Interventions: Drug: Fentanyl Injection

INTERVENTIONS:
Drug: Fentanyl infusion — will received lidocaine with dose 250 mg and fentanyl infusion in dose of 200 µg in rate 10ml /hr using 50ml syringe pump.
  Arms: group 1
Drug: Fentanyl Injection — will receive lidocaine 250 mg in addition to fentanyl injection in dose 100 µg by shots
  Arms: group 2

SUMMARY:
Injury and deformity of the upper extremity can result in dysfunction to nerves, tendons and bones which can lead to disability and pain.

Various techniques of regional anesthesia are frequently used for upper extremity surgery. Specifically, intravenous regional anesthesia, the Bier block, is an effective anesthetic technique. This technique, developed by Dr August Bier in 1908, provides complete anesthesia, a bloodless field, and eliminates the need for general anesthesia. However, it was not until the 1960s that this technique was reintroduced and used in upper extremity surgery due to several disadvantages and reports of major complications. Because of the dose of lidocaine and tourniquet time, there is potential for cardiac and neurological complications such as arrhythmias, seizures, and compartment syndrome the aim of this study To evaluate the effect of Systemic Fentanyl Infusion compared to addition of Fentanyl as An Adjuvant to Lidocaine in Bier Block for Controlling Pain in Patients Undergoing Hand Surgeries

DETAILED DESCRIPTION:
Injury and deformity of the upper extremity can result in dysfunction to nerves, tendons and bones which can lead to disability and pain.

Various techniques of regional anesthesia are frequently used for upper extremity surgery. Specifically, intravenous regional anesthesia, the Bier block, is an effective anesthetic technique. This technique, developed by Dr August Bier in 1908, provides complete anesthesia, a bloodless field, and eliminates the need for general anesthesia. However, it was not until the 1960s that this technique was reintroduced and used in upper extremity surgery due to several disadvantages and reports of major complications. Because of the dose of lidocaine and tourniquet time, there is potential for cardiac and neurological complications such as arrhythmias, seizures, and compartment syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients age from 18 years to 40 years

  * Both sex
  * Patients of the American Society of Anesthesiologists (ASA) physical Status class I and II
  * BMI less than 40

Exclusion Criteria:

* • Patients who refuse to participate in study.

  * Uncooperative patients.
  * Patient with crush injury
  * Peripheral vascular, neurological or muscle diseases.
  * Coagulation disorders that affect the blood's clotting activities e.g.: Hemophilia.
  * History of hypersensitivity to the drugs being evaluated

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
to compare intraoperative pain between systemic and local fentanyl using VAS score | baseline
  pain will be assessed using an 11-point (0=no pain and 10=worst pain) VAS scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jung H, Lee KH, Jeong Y, Lee KH, Yoon S, Kim WH, Lee HJ. Effect of Fentanyl-Based Intravenous Patient-Controlled Analgesia with and without Basal Infusion on Postoperative Opioid Consumption and Opioid-Related Side Effects: A Retrospective Cohort Study. J Pain Res. 2020 Nov 24;13:3095-3106. doi: 10.2147/JPR.S281041. eCollection 2020. PMID 33262644
- [Background] Glick JL, Christensen T, Park JN, McKenzie M, Green TC, Sherman SG. Stakeholder perspectives on implementing fentanyl drug checking: Results from a multi-site study. Drug Alcohol Depend. 2019 Jan 1;194:527-532. doi: 10.1016/j.drugalcdep.2018.10.017. Epub 2018 Nov 13. PMID 30551090
- [Background] Farzam R, Deilami M, Jalili S, Kamali K. Comparison of Anesthesia Results between Wide Awake Local Anesthesia no Tourniquet (WALANT) and Forearm Tourniquet Bier Block in Hand Surgeries: A Randomized Clinical Trial. Arch Bone Jt Surg. 2021 Jan;9(1):116-121. doi: 10.22038/abjs.2020.49526.2487. PMID 33778124
- [Background] Badeaux J, Bonanno L, Au H. Effectiveness of ondansetron as an adjunct to lidocaine intravenous regional anesthesia on tourniquet pain and postoperative pain in patients undergoing elective hand surgery: a systematic review protocol. JBI Database System Rev Implement Rep. 2015 Jan;13(1):27-38. doi: 10.11124/jbisrir-2015-1768. PMID 26447005